CLINICAL TRIAL: NCT06679699
Title: "Effectiveness of Patient Education Program About Trunk Control Exercises on Balance and Functional Mobility in Individuals With Post-stroke Hemiparesis: A Randomized Control Trial"
Brief Title: Patient Education Program and Trunk Control Exercises in Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-09-DEC-2020
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Strokes Thrombotic
Keywords: Stroke; Hemiparesis; Trunk control; Patient education; Balance
MeSH Terms: conditions — Thrombotic Stroke; Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was blinded to the participants allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk control exercises with Patient education program (Experimental): This group have received Trunk control exercises along with patient education program.
  Interventions: Device: Trunk control exercises combined with patient education program
- Trunk control exercises (Active Comparator): This group have received standalone trunk control exercises.
  Interventions: Device: Trunk control exercises

INTERVENTIONS:
Device: Trunk control exercises combined with patient education program — Patients in this group received about 45-60 minutes of trunk control exercises in lying and sitting, 5 days a week for 4 consecutive weeks. Each exercise was performed with 10-20 repetitions per session depending on the patient's ability. Trunk exercises or other activities targeting the trunk while sitting and lying, to minimize the influence of lower extremity function performed either on a stable or unstable surfaces. In addition, the experimental group provided a patient education program which focuses on the importance of trunk control and benefits of trunk control exercises during the rehabilitation process. Further, caregivers and family members were also explained about the patient education program and adherence with treatment protocol during and after the interventions.
  Arms: Trunk control exercises with Patient education program
Device: Trunk control exercises — Patients in this group received about 45-60 minutes of trunk control exercises in lying and sitting, 5 days a week for 4 consecutive weeks. Each exercise was performed with 10-20 repetitions per session depending on the patient's ability. Trunk exercises or other activities targeting the trunk while sitting and lying, to minimize the influence of lower extremity function performed either on a stable or unstable surfaces.
  Arms: Trunk control exercises

SUMMARY:
The trunk movement awareness and education of individuals with post-stroke hemiparesis is not emphasized adequately in clinical practice. Therefore, this current study was made to hypothesize whether a patient education program about dynamic trunk control exercises during stroke rehabilitation may influence trunk control. 40 individuals with post-stroke hemiparesis were recruited and randomly allocated to the experimental and control group. Both the groups received 1 hour of exercises focusing more on dynamic trunk control exercises with patient education chart (experimental group) and without the patient education chart (control group) for 4 weeks.

DETAILED DESCRIPTION:
The prevalence of stroke in adults increased by 14.6% in 2022 compared to data collected in 2013. Poor balance, postural asymmetry, abnormal gait, and fall-related complications due to reduced trunk control can limit social interactions. Trunk control is an important predictor of functional independence for stroke-affected individuals recovering from functional impairments. Studies have found that individuals with post-stroke hemiparesis have mild-to-severe trunk dysfunction even 6 months post-stroke occurrence. Evidence also indicates that the muscular strength of the trunk is significantly reduced in acute and chronic stages, which leads to poor functional performance. As trunk function significantly contributes to functional recovery, the importance of trunk training needs to be emphasized, and education should be provided to stroke patients for faster functional mobility.

Patient education programs guide patients, caregivers, and family members to understand and promote the patient's participation in continuing care and treatment decisions. This method assists patients in incorporating information, expertise, beliefs, and behaviors related to their health promotion and faster functional recovery from physical and psychological impairments. Patient education provides adequate and appropriate scientific knowledge for patients to improve their awareness of illness conditions and health-promoting practices. Studies also suggest that the patient education process increases patient's involvement in rehabilitation practices.

Although trunk control exercises are performed during routine rehabilitation programs, knowledge and education about trunk training exercises are not specifically emphasized in stroke rehabilitation protocols. Stroke patients need to be educated not only about upper and lower functional training but also should understand trunk control training during their rehabilitation process to acquire skills.

In this proposed study, a patient education program highlighting the significance of trunk control, its role in functional improvement, and patient-centered self-care might provide better functional mobility compared to a standalone trunk control exercises program. Through this program, patients can concentrate not only on limb training but also emphasize trunk-related functional tasks to improve overall body function. Therefore, our current study hypothesized that a patient education program about the trunk training program during the rehabilitation process may improve balance and functional mobility better than a standalone trunk control exercises program in patients with post-stroke hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ischemic stroke
* Grade 1 - 2 Spasticity
* Hemiparesis

Exclusion Criteria:

* Moderate to severe cognitive deficits,
* Alzheimer's disease,
* Language difficulties,
* Unstable blood pressure
* Uncontrolled epilepsy,
* Dislocations/fractures

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Trunk impairment scale | Baseline, post-treatment week 4
  The Trunk Impairment Scale (TIS) is a valid tool for assessing motor impairment of the trunk in stroke patients. In a sitting position, patient's static and dynamic sitting balance, as well as trunk coordination were assessed. For the static subscale, the patient's ability to maintain a sitting position with feet supported and legs crossed. The lateral flexion of the trunk and unilateral hip lifting were assessed to quantify the dynamic sitting balance. To assess the coordination function, the patient was instructed to rotate the upper or lower part of their trunk six times, initiating movements from the shoulder or pelvic girdle. The total score ranges from 0 (minimal performance) to 23 (perfect performance). This scale has high reliability, validity, and predictive value for functional outcomes, making it an effective tool for evaluating trunk function in stroke patients

SECONDARY OUTCOMES:
Functional Mobility | Baseline, post-treatment week 4
  The Rivermead Mobility Index (RMI) is a valid tool for assessing functional mobility in stroke patients. It is the 15-item questionnaire, which includes 14 self-reported items and one direct observation task. The items cover a range of mobility activities, from turning in bed to running. For each item, the patient receives a score of 1 if they can perform the task independently, or 0 if they cannot. The assessor allowed the patient to attempt each task unless there is a safety concern. The total score ranges from 0 to 15, with higher scores indicating better functional mobility
Berg Balance Scale | Baseline, post-treatment week 4
  The Berg Balance Scale (BBS) is a valid and reliable tool, consisting of 14-items that evaluates a patient's ability to maintain balance while performing functional tasks. The assessment items range from simple activities like sitting unsupported to more challenging tasks such as standing on one foot. Each item is scored on a 5-point ordinal scale from 0 (unable to perform) to 4 (independent) depending on the patient's achievement level. A score of ≤49/56 indicates a fall risk in stroke patients and change of 4-7 points considered clinically significant improvement

CONTACTS AND LOCATIONS:
Overall Officials: Ramprasad Muthukrishnan, PDF, Study Chair — Gulf Medical University
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
The data may be provided based upon request related to research purpose